CLINICAL TRIAL: NCT06947122
Title: Mindfulness-Based Ecological Momentary Intervention for Co-Occurring Opioid Use Disorder and Chronic Pain: A Pilot Study
Brief Title: Mindfulness-Based Ecological Momentary Intervention for Opioid Use Disorder and Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Chung Jung Mun, Associate Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019109
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Opioid Use Disorder
Keywords: mindfulness; opioid use disorder; chronic pain; mHealth; ecological momentary intervention
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluating the Feasibility and Acceptability of Mindful Journey Prototype (Experimental): In this single arm trial, participants will complete surveys and interviews about experiences with opioid and other substance use, chronic pain, and treatments, and a brief timeline follow-back assessment for substance use. Participants will also be completing a training session to learn about the study procedure, and the mobile app platform. Participants will enter the intervention period (8-weeks) and complete 14 foundational modules throughout the intervention period using the Mindful Journey app. Daily brief check-in surveys will be completed via the app. Based on these survey responses, participants will receive brief, tailored momentary mindfulness coaching. Study staff will also conduct weekly phone check-ins to support engagement. The final visit will occur following the intervention period and the participant will complete a series of self-report batteries and participate in a brief exit interview to gather feedback and suggestions for improving the app.
  Interventions: Behavioral: Mindfulness based smartphone app

INTERVENTIONS:
Behavioral: Mindfulness based smartphone app — The Mindful Journey intervention includes (1) 14 foundational modules/lessons, (2) brief check-in surveys (3 times/day) via the app, (3) app-guided momentary mindfulness coaching (max 3 times/day), and (4) brief phone-based check-in from a trained staff member, on a weekly basis. Occurring for approximately 8 weeks following enrollment visit
  Other Names: Mindful Journey

SUMMARY:
The goal of this clinical trial is to evaluate whether a smartphone app-based ecological momentary intervention called Mindful Journey, which teaches mindfulness skills, can support adults in recovery from both opioid use disorder and chronic pain. The primary objective of this pilot study is to assess the feasibility and acceptability of Mindful Journey in this population.

DETAILED DESCRIPTION:
There is a paucity of interventions for co-occurring opioid use disorder and chronic pain. Difficulty with emotion regulation is a key shared vulnerability factor underlying both conditions. Mindfulness-Based Interventions (MBIs) are a promising intervention approach, as they target core skills that can improve emotion regulation. However, research on MBIs for co-morbid opioid use disorder and chronic pain is limited. Existing MBIs are also limited by not providing adequate support "in the moment" when individuals are in high-risk situations. A responsive, momentary MBI for co-occurring opioid use disorder and chronic pain may be highly promising, but has yet to be established. In the present study, we will be evaluating a smartphone app-based ecological momentary intervention, called Mindful Journey, for individuals with opioid use disorder and chronic pain. The core feature of the app is training in mindful acceptance and savoring skills via momentary "just-in-time" delivery of brief video-based exercises based upon ecological momentary assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* fluent in English
* enrollment in medication-assisted treatment for opioid use disorder
* report at least bothersome chronic pain, as indicated by Graded Chronic Pain Scale-Revised
* has a smartphone.

Exclusion Criteria:

* self-reporting of chronic malignant pain (e.g., cancer) or systemic inflammatory disease (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus, and sarcoidosis)
* self-reporting of psychotic disorder symptoms
* participated in the previous phase of the study in which participants provided feedback to inform the development of the Mindful Journey app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dimensions of acceptability of the Mindful Journey lessons | Assessed at the end of the 8-week treatment period
  Single-items measuring ratings of acceptability dimensions for the lessons, including usability, understandability, engage-ability, visual appeal, helpfulness, skill acquisition, and confidence implementing skills. Scores for each item range from 1 to 5, with higher scores indicating better acceptability.
Dimensions of acceptability of the ecological momentary intervention (momentary coaching) | Assessed at the end of the 8-week treatment period
  Single-items measuring ratings of acceptability dimensions for ecological momentary intervention (momentary coaching), including usability, understandability, engage-ability, visual appeal, helpfulness, skill acquisition, and confidence implementing skills. Scores for each item range from 1 to 5, with higher scores indicating better acceptability.
Momentary ratings of acceptability of the ecological momentary intervention (momentary coaching) | Administered immediately after participants receive each ecological momentary intervention (momentary coaching)
  Single item of perceived helpfulness
Completion rates for the lessons on the Mindful Journey | 8-week treatment period
  Percent of lessons completed
Completion rates for ecological momentary intervention (momentary coaching) | 8-week treatment period
  Percent of ecological momentary interventions (momentary coaching) completed
Completion rates for momentary check-in surveys | 8-week treatment period
  Percent of momentary check-in surveys completed

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Phoenix, Arizona
  - Arizona State University Downtown Phoenix Campus, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the primary goal of this pilot study is to assess feasibility and acceptability, not to generate generalizable efficacy data suitable for secondary analyses.

REFERENCES:
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Von Korff M, DeBar LL, Krebs EE, Kerns RD, Deyo RA, Keefe FJ. Graded chronic pain scale revised: mild, bothersome, and high-impact chronic pain. Pain. 2020 Mar;161(3):651-661. doi: 10.1097/j.pain.0000000000001758. PMID 31764390
- [Background] Wong SYS, Chan JYC, Zhang D, Lee EKP, Tsoi KKF. The safety of mindfulness-based interventions: a systematic review of randomized controlled trials. Mindfulness (N Y). 2018;9:1344-1357.